CLINICAL TRIAL: NCT02568748
Title: Evaluation of Cytokine-induced Killer (CIK) Cells as Therapy or Adjuvant Treatment for Patients With Advanced Hepatocelluler Carcinoma
Brief Title: Evaluation of Cytokine-induced Killer (CIK) Cells as Therapy or Adjuvant Treatment for Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Study director, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIK Tanta university
Record Dates: First submitted 2015-10-04; First posted 2015-10-06 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CIK with TACE for HCC stage B (Experimental): HCC patients stage B treated with TACE and CIK as adjuvant therapy.
  Interventions: Biological: CIK; Procedure: TACE
- TACE only for HCC stage B (Experimental): HCC patients stage B treated with TACE without receiving CIK cells infusion
  Interventions: Procedure: TACE
- CIK in HCC stage C or D (Experimental): HCC stage C or D will receive supportive treatment in addition to CIK cells infusion
  Interventions: Biological: CIK
- Supportive treatment in HCC stage C or D (No Intervention): HCC stage C or D will receive supportive treatment only .

INTERVENTIONS:
Biological: CIK — Cytokine -induced killer cells in Egyptian patients with advanced hepatocellular carcinoma as treatment or adjuvant treatment in comparison with traditional treatment.
  Arms: CIK in HCC stage C or D; CIK with TACE for HCC stage B
Procedure: TACE — Trans-arterial chemoembolization
  Arms: CIK with TACE for HCC stage B; TACE only for HCC stage B

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common malignancy in the world and the third most common cause of cancer-related deaths complicating liver cirrhosis in most cases. In Egypt, there has been a remarkable increase of the proportion of HCC among CLD patients from 4.0% to 7.2% over a decade. This rising proportion may be explained by the increasing risk factors such as the emergence of HCV over the same period of time, the contribution of HBV infection, improvement of the screening programs and diagnostic tools of HCC as well as the increased survival rate among patients with cirrhosis to allow time for some of them to develop HCC. The only curative treatment modalities for HCC are surgery, local ablation, and liver transplantation which have high recurrence rate either due to viral hepatitis infection or cirrhosis leading to low success rate and high economic burden.

Unfortunately, the majority of patients have unresectable disease at diagnosis. So, patients search for palliative very expensive therapies including chemotherapy and radiotherapy which often fail to eradicate tumor lesions completely and tend to result in many adverse events.Thus, novel approaches for treatment options are needed for patients with advanced HCC .

In recent years, immunotherapy has emerged as an efficacious treatment modality with encouraging efficacy and slight adverse events in cancer therapy [Stroncek 2010]. Cytokine-induced killer CIK cells therapy has been evaluated as an adoptive cell immunotherapy for cancer patients in a number of clinical trials and the promising efficacy of CIK cells on malignancies has been proved.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common malignancy in the world and the third most common cause of cancer-related deaths complicating liver cirrhosis in most cases. In Egypt, there has been a remarkable increase of the proportion of HCC among CLD patients from 4.0% to 7.2% over a decade. This rising proportion may be explained by the increasing risk factors such as the emergence of HCV over the same period of time, the contribution of HBV infection, improvement of the screening programs and diagnostic tools of HCC as well as the increased survival rate among patients with cirrhosis to allow time for some of them to develop HCC. The only curative treatment modalities for HCC are surgery, local ablation, and liver transplantation which have high recurrence rate either due to viral hepatitis infection or cirrhosis leading to low success rate and high economic burden..

Unfortunately, the majority of patients have unresectable disease at diagnosis. So, patients search for palliative very expensive therapies including chemotherapy and radiotherapy which often fail to eradicate tumor lesions completely and tend to result in many adverse events.Thus, novel approaches for treatment options are needed for patients with advanced HCC .

In recent years, immunotherapy has emerged as an efficacious treatment modality with encouraging efficacy and slight adverse events in cancer therapy. Cytokine-induced killer CIK cells therapy has been evaluated as an adoptive cell immunotherapy for cancer patients in a number of clinical trials and the promising efficacy of CIK cells on malignancies has been proved. . Clinical studies have demonstrated that it is an excellent method to prevent tumor recurrence and has preliminarily shown its efficacy in inhibiting recurrence and metastasis of primary HCC -Peripheral blood mononuclear cells (PBMC)from patients with primary HCC were incubated in vitro and induced into CIK cells in the presence of various cytokines such as interferon-gamma (IFN-ã ), interleukin-1 (IL-1), IL-2, and monoclonal antibody (mAb) against CD3. CIK cells infusion will be performed Once every week, with a total of at least4infusions. Infusion will be given intrahepatic or via peripheral veins .

The serial biological events following CIK cells administration to a cancer patient includes (a) immune activation and effective lymphocytes (mostly C D3+CD 5 6+Tlymphocytes) proliferation starting early after the first administration , ( b) clinically measurable antitumor effect mediated by activated immune cells over weeks to months ,and (c) potential delayed effect on patient survival several months or even longer after the first administration.

Our team have many grants in field of HCC biomarkers discovery and managements from NIH as multicenter studies which got many international publication. As well as grant for the use of laboratory techniques in the cultivation of stem cells for specialized cells used in the treatment of different diseases which got publication in this era. we aim in this project to cultivate patients cells in vitro to get CIK cells and study the safety and efficacy of immunization with specific antihepatocellular carcinoma Cytokine -induced killer cells in Egyptian patients with advanced hepatocellular carcinoma as treatment or adjuvant treatment in comparison with traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced HCC and not fit for resection or local ablative therapies stage B (according Barcelona Clinic Liver Cancer (BCLC) Staging system ).
2. Patient with HCC and portal vein thrombosis stage C.
3. Patients with HCC and lymphatic or distant metastases stage D.

Exclusion Criteria:

1. Patients with HCC and fit for radical or local ablation (stage 0 and A) therapies.
2. Platelet count below 50,000 / dl
3. Prothrombin activity below 50%
4. All patients will sign a written informed consent after explaining the details and possible hazards of the procedure to them. Those who will refuse to share in the study will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with ablated hcc | 1 year
  patients with ablated hcc

CONTACTS AND LOCATIONS:
Overall Officials: Dina H Ziada, Prof, Principal Investigator — Hepatology dept.-Tanta; Hanan H Soliman, Prof, Study Director — Hepatology dept.-Tanta; Enas Arafa, Prof, Study Director — Clinical pathology dept.; Sherief Abd-Elsalam, lecturer, Study Director — Hepatology dept.-Tanta; Abdelrahman Zekri, Professor, Study Chair — Pathology dept.- Cairo university; Amre Elbadry, Professor, Study Chair — Interventional radiology- Tanta university; Marwa Salama, Ass.lecturer, Study Chair — Hepatology dept.- Tantauniversity; Ahmed Elsharkawy, Ass.lecturer, Study Chair — Interventional radiology- Tanta university
Locations (1):
- Sherief Abd-Elsalam, Cairo, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided